CLINICAL TRIAL: NCT01215747
Title: International Randomized, Double-Blind, Placebo-Controlled, Phase 3 Study of the Efficacy and Safety of KIACTA in Preventing Renal Function Decline in Patients With AA Amyloidosis
Brief Title: Efficacy and Safety Study of KIACTA in Preventing Renal Function Decline in AA Amyloidosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: C.T. Development America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CL-503012
Record Dates: First submitted 2010-10-01; First posted 2010-10-06 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-03

CONDITIONS: Amyloidosis
Keywords: Kiacta for AA amyloidosis
MeSH Terms: conditions — Amyloidosis | interventions — eprodisate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Kiacta (eprodisate disodium) (Experimental)
  Interventions: Drug: KIACTA (eprodisate disodium)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: KIACTA (eprodisate disodium) — Orally 1 to 3 capsules (Kiacta 400 mg) twice daily and adjusted as per the Creatine Clearance (CrCl) level increases or decreases.
  Arms: Kiacta (eprodisate disodium)
Drug: Placebo — Orally 1 to 3 capsules (placebo) twice daily and adjusted as per the Creatine Clearance (CrCl) level increases or decreases:
  Arms: Placebo

SUMMARY:
The primary purpose of this study is to assess the efficacy and safety of treatment with Kiacta in adult patients with AA Amyloidosis.

ELIGIBILITY:
Inclusion Criteria:

* females must be of nonchildbearing potential (more than 1 yr postmenopausal)or use effective contraception for at least 2 months prior to the baseline visit and through 30 days after the last dose of study medication
* confirmed diagnosis of AA amyloidosis demonstrated by positive biopsy using congo red staining and immunohistochemistry or immunoelectronmicroscopy. Mass spectroscopy will be used upon approval of the sponsor on a case to case basis.
* persistent proteinuria greater than 1 g/24h at 2 distinct 24-hr urine collections
* must have CrCl greater than 25 ml/min/1.73 m2 at 2 distinct 24 hr urine collections

Exclusion Criteria:

* evidence or suspicion of chronic kidney disease secondary to a disease other than AA amyloidosis (eg, diabetes, long-standing uncontrolled hypertension, polycystic kidney disease, recurring polynephritis, or systemic lupus erythematosus)
* history of kidney transplantation
* evidence or suspicion of a cause of potentially reversible acute renal failure within 3 months prior to baseline visit
* presence of concomitant diseases or medication that could interfere with the interpretation of study results or compromise patient safety
* presence of condition that could reduce life expectancy to less than 2 yrs
* Type 1 or 2 diabetes mellitus
* significant hepatic enzyme elevation
* unstable angina, myocardial infarction, coronary artery bypass graft surgery, or percutaneous transluminal coronary angioplasty within 6 months prior to the baseline visit; presence of NY Heart Assoc class III or IV heart failure
* presence of, or history of stroke or transient ischemic attack within 6 months prior to baseline visit
* initiation of, or any changes in, angiotensin converting enzyme inhibitor, angiotensin II receptor antagonist therapy, or renin inhibitor within 3 months prior to baseline visit
* initiation of, or any changes in, cytotoxic agents, anti-tumor necrosis factor agents, anti interleukin-1 or 6 agents, or colchicine therapy within 3 months prior to baseline visit
* previous use of Kiacta
* history of malignancy within 5 yrs prior to study entry, except for cervical carcinoma in situ, nonmelanomatous carcinoma of the skin, or ductal carcinoma in situ of the breast that has been surgically cured
* use of investigational drug within 30 days prior to the first screening visit
* active alcohol and/or drug abuse

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 261 (Actual)
Dates: Start 2010-11; Primary Completion 2016-01 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Time from baseline to a persistent decrease in Creatinine clearance (CrCL) of 40% or more, a persistent increase in Serum Creatinine(SCr) of 80% or more, or progression to end-stage renal disease(ESRD) | Up to 24 months

SECONDARY OUTCOMES:
rate of change (slope) in creatinine clearance (CrCL) over time | baseline to primary endpoint, measured every 3 months to end of study visit
Progression to end-stage renal disease (ESRD) | baseline, every 3 months to end of study visit
estimated glomerular filtration rate (eGFR) | screening, baseline, every 3 months, 12 months , early termination, treatment completion, end of study visit
serum cystatin C over time | baseline, every 3 months, 12 months, early termination, treatment completion, end of study visit
urinary protein/creatinine ratio | screening, baseline, every 3 months, 12 months, early termination, treatment completion, end of study visit
serum amyloid A | baseline, every 3 months, 12 months, early termination, treatment completion, end of study visit
Time from baseline to persistent decrease in CrCL of 40% or more, a persistent increase in SCr of 80% or more, progression to ESRD, or all-cause mortality | Up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Sablinski, MD, PhD, Study Director — CT Development America, Inc.
Locations (45):
- United States (3):
  - Raffi Minasian MD a Medical Corporation, Glendale, California
  - Boston Medical Center, Boston, Massachusetts
  - Ohio State University Medical Center, Columbus, Ohio
- UZ Leuven, Leuven, Belgium
- Al Hussain University Hospital, Cairo, Egypt
- Tartu University Hospital, Tartu, Estonia
- Helsingin yliopistollinen keskussairaala / Meilahti, Helsinki, Finland
- France (2):
  - Hôpital Henri Mondor, Créteil
  - Hôpital Claude Huriez, Lille
- Tbilisi Heart and Vascular Clinic Ltd, Tbilisi, Georgia
- Universität Heidelberg, Heidelberg, Germany
- India (3):
  - Regency Hospital, Kanpur
  - Muljibhai Patel Urological Hospital, Nadiād
  - Sir Ganga Ram Hospital, New Delhi
- Israel (2):
  - Bnei Zion Medical Center, Haifa
  - The Chaim Sheba Medical Center, Ramat Gan
- IRCCS Policlinico San Matteo, Pavia, Italy
- Pauls Stradins Clinical University Hospital, Riga, Latvia
- Lithuania (2):
  - Hospital of Lithuanian University of Health Sciences Kaunas Clinics, Kaunas
  - Vilnius University Hospital Santariskiu Klinikos, Vilnius
- Netherlands (2):
  - Universitair Medisch Centrum Groningen, Groningen
  - Academisch Ziekenhuis Maastricht, Maastricht
- Hospital Nacional Arzobispo Loayza, Lima, Peru
- Poland (3):
  - Wojewodzki Szpital Specjalistyczny, Olsztyn
  - ARS RHEUMATICA Sp. z o.o., Warsaw
  - Akademicki Szpital Kliniczny im. Jana Mikulicza-Radeckiego we Wroclawiu, Wroclaw
- Russia (4):
  - Kemerovo State Medical Academy of Roszdrav, Kemerovo
  - Institute of Rheumatology of RAMN, Moscow
  - Research Institute of Clinical and Experimental Lymphology, Novosibirsk
  - Sverdlovsk Regional Clinical Hospital #1, Yekaterinburg
- Spain (2):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Civil Carlos Haya, Málaga
- Karolinska Universitetssjukhuset i Huddinge, Stockholm, Sweden
- Tunisia (5):
  - Fattouma Bourguiba University Hospital, Monastir
  - Hedi Chaker University Hospital, Sfax
  - Sahloul Hospital, Sousse
  - Hôpital Charles Nicolle, Tunis
  - La Rabta Hospital, Tunis
- Turkey (Türkiye) (3):
  - Cukurova University Medical Faculty Balcali Hospital, Adana
  - Hacettepe University Medical Faculty, Ankara
  - Eskisehir Osmangazi University Medical Faculty, Eskişehir
- Ukraine (3):
  - Municipal Medical & Preventive Institution Donetsk Regional Clinical Territorial Medical Association, Donetsk
  - National Scientific Center "Institute of cardiology n.a. academician M.D Strazhesko", Kyiv
  - State Institution "Institute of Nephrology of AMS of Ukraine", Kyiv
- Royal Free Hospital, London, United Kingdom